CLINICAL TRIAL: NCT00550914
Title: A Multi-Center, Randomized, Controlled Trial of the Pulsed Dye Laser for Juvenile Onset Recurrent Respiratory Papillomatosis
Brief Title: Multi-Center, Randomized Trial of the Pulsed Dye Laser for JORRP
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Christopher Hartnick, M.D., Principal Investigator, Massachusetts Eye and Ear Infirmary
Other Study IDs: 07-01-005; 07-01-005
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: Papilloma, Papillomatosis, Laser, Laser Surgery
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Papilloma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control arm: The conventional therapy arm will undergo debridement with either a powered microdebrider or cold instrumentation excision as per the preference of the individual surgeon. Debridement will be deemed complete after removal of gross papilloma to the extent that the individual surgeon feels can be safely accomplished. Standard microsurgical principles of the larynx will guide debridement in that no opposing mucosal surfaces of the true vocal folds, laryngeal ventricle or inter-arytenoid space will be simultaneously debrided
- Experimental Arm: Patients enrolled into the conventional therapy plus PDL treatment arm will undergo debridement of the supraglottis and subglottis via conventional techniques as per the individual surgeons preferences followed by therapy to anterior commissure, true vocal folds, laryngeal ventricle and inter-arytenoid space with the pulsed dye laser. Standard laser settings will be a 450 microsecond pulse width, 5 J per pulse maximum of 1Hz, 1 mm spot fiber, 1-2 mm spot size and fluences of 38-255 J/cm2.

SUMMARY:
The purpose of this study is to determine whether the 585-nm pulse dye laser can decrease the time interval between surgeries and improve voice outcomes in children with severe RRP.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompetent children ages 1-12 with symptomatic JORRP requiring operative intervention
2. Children who have historically required at least four surgeries in the year preceding enrollment to treat laryngeal JORRP

Exclusion Criteria:

1. Children who have required fewer than four procedures to treat laryngeal JORRP in the year prior to enrollment.
2. Children who are currently receiving adjuvant therapies for JORRP including cidofovir, interferon, indole-3-carbinol or Hsp-E7.
3. Caregivers who are non-English speaking as the PVRQOL instrument has been validated only in the English language.
4. Children whose families do not sign an informed consent to enter into the study.
5. Children whose families anticipate discontinuing care at a participating institution during the study period

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with severe JORRP
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2007-01; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Measure: Time interval between surgical therapy for recurrent respiratory papillomatosis | One Year

SECONDARY OUTCOMES:
Measure: Validated voice questionnaire and intraoperative laryngoscopic staging score | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hartnick, M.D., Study Chair — Massachusetts Eye and Ear Infirmary
Locations (2):
- United States (2):
  - Rady Children's Hospital, San Diego, California
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts